CLINICAL TRIAL: NCT03690024
Title: Outcame of Cases With Hemolytic Uremic Syndrome Attending Assiut University Child Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, walaa gamal abd elrazik, Principal investigator, Assiut University
Other Study IDs: Ocwhus
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Hemolytic Uremic Syndrome of Childhood

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diarrhea-associated hemolytic uremic syndrome (D+HUS) is defined as a prodrome of enteritis followed by thrombocytopenia (< 150,000/mm3), microangiopathic hemolytic anemia, and signs of variable degrees of renal damage (increase in serum Cr, proteinuria, and/or hematuria) . Our aim is to detect the most reliable early predictors of poor prognosis to identify children at major risk of bad outcome who could eventually benefit from early specific treatments.

DETAILED DESCRIPTION:
The disease is caused predominantly by Shiga toxin-producing enterohemorrhagic Escherichia coli (STEC) and is one of the most common etiologies of acute kidney injury (AKI) and an important cause of acquired chronic kidney disease in children [2]. The incidence of HUC tends to parallel the seasonal fluctuation of E.coli o175 : H7 infection which peaks between June & September. Nowadays, the incidence increases and is typically observe in infants and children, especially those aged 6 months to 4 years. A complicated disease course is defined as the development of one or more of the following manifestations: neurological dysfunction, severe bowel injury, pancreatitis, hemodynamic instability (symptomatic hypotension, multi-organ failure), cardiac (congestive heart failure, myocarditis, pericarditis, arrhythmia) or pulmonary involvement (pulmonary edema, acute respiratory distress syndrome), hematologic complications (hemorrhage), and death [1].

Many laboratory and clinical markers upon admission have been associated to severe forms of the disease, including high initial leukocyte and hematocrit levels, major extrarenal complications, dehydration and recently, the blood urea nitrogen (BUN) to serum creatinine (Cr) ratio [1], [4-6]. Treatment of D+HUS remains supportive; thus, early identification of high-risk patients can optimize their management [1-3].

ELIGIBILITY:
Inclusion Criteria:

* all patients less than 18 years diagnosed with Hemolytic Uremic Syndrome

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients attending Assiut University Child hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 1 year
  Number of cases that treated and discharged from hospital
Death | 1 year
  Number of cases that ended by death
Residual renal affection | 1 year
  Number of cases with residual raised renal chemistry